CLINICAL TRIAL: NCT01651767
Title: A Phase Ib, Randomized, Double-Blind, Placebo-Controlled Trial in Caucasian Genotype 1 Chronic HCV-Infected Subjects to Determine the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Repeated Doses of JNJ-47910382 Given in Different Doses and Dose Regimens
Brief Title: Study in HCV-Infected Patients to Determine the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of JNJ-47910382
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Because of many competing trials using the same mechanism of action, but being further advanced in development
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR100760; 47910382HPC1002 (Other: Janssen R&D Ireland); 2011-005110-10 (EudraCT Number)
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Chronic hepatitis C virus infection; JNJ-47910382; Pharmacokinetics; Caucasian genotype-1; Non-structural protein 5A (NS5A) inhibitor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Panel I (Experimental): Patients will be randomized to receive JNJ-47910382 at a dose of 30 mg or placebo as monotherapy once daily for 5 days.
  Interventions: Drug: Placebo; Drug: JNJ-47910382
- Panel II (Experimental): Patients will be randomized to receive JNJ-47910382 at a dose of 90 mg or placebo as monotherapy once daily for 5 days.
  Interventions: Drug: Placebo; Drug: JNJ-47910382
- Panel III (Experimental): Patients will be randomized to receive JNJ-47910382 at a dose of 300 mg or placebo as monotherapy once daily for 5 days.
  Interventions: Drug: Placebo; Drug: JNJ-47910382
- Panel IV (Experimental): Patients will be randomized to receive JNJ-47910382 at a dose of 400 or 450 mg once daily or 300 mg twice daily (morning dose only on Day 5) or placebo as monotherapy for 5 days.
  Interventions: Drug: Placebo; Drug: JNJ-47910382

INTERVENTIONS:
Drug: Placebo — Form=suspension, route=oral.
Drug: JNJ-47910382 — Type=exact number, unit=mg, number=30, 90, 300, 400 or 450, form=suspension, route=oral. Study drug will be administered once or twice daily

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics (what the body does to the medication) and antiviral activity of JNJ-47910382 when administered in different dosing regimens in Caucasian genotype-1 chronic HCV-infected patients.

DETAILED DESCRIPTION:
This is a Phase Ib, double-blind (neither physician nor patient knows the treatment that the patient receives), randomized (the study drug is assigned by chance), placebo-controlled study in treatment-naïve (someone who has never used drugs for HCV infection), Caucasian genotype 1 chronic HCV-infected patients. The study consists of a screening period, a 9-day treatment period (with 5 days of actual medication intake) and a 4-week follow-up period. The patients will be divided over 4 panels of 10 patients each that will be initiated sequentially. In each panel patients will receive JNJ-47910382 or placebo during 5 consecutive days. JNJ-47910382 or placebo will be administered once daily or twice daily. Within each panel, 5 patients of genotype-1a and 5 patients of genotype-1b will be enrolled. Patients will be randomly assigned to receive active treatment or placebo in such a way that 4 patients of each genotype receive active treatment and 1 subject of each genotype receives placebo. The pharmacokinetic profile of JNJ-47910382 will be assessed in each panel. HCV RNA kinetics (HCV RNA level) and HCV resistance will be studied and biomarkers at the messenger RNA (mRNA), protein and cell level will be explored. The entire study duration for each participant will be approximately four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (diagnosis of hepatitis C more than or 6 months before the screening period) HCV infection. Geno- and subtype should be determined or confirmed at screening, and should be 1a or 1b
* Never received (Peg) IFN, RBV or any other approved or investigational antiviral treatment for chronic HCV infection
* HCV RNA level of >100,000 IU/mL at screening (as assessed by standard quantitative in vitro nucleic acid amplification assay)
* Patients having good accessible veins

Exclusion Criteria:

* Evidence of liver cirrhosis or decompensated liver disease
* Patient coinfected with HIV-1 or HIV-2, or hepatitis A or B virus infection, or active tuberculosis at study screening
* Patient infected/coinfected with non-genotype-1 HCV at study screening
* Patient with any cardiac disease at screening, or any active clinically significant disease, or medical history or physical examination findings during screening
* Patient having uncontrolled/unstable disease such as diabetes, epilepsy, a manifest psychiatric disease, thyroid disease or disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Determination of pharmacokinetics of JNJ-47910382 | Up to 9 Days
  The pharmacokinetics of JNJ-47910382 after 5 consecutive days of administration in chronic HCV-genotype-1 infected patients in different doses and dose regimens will be determined.
Evaluation of the intrinsic antiviral activity of JNJ-47910382 | Up to 4 weeks
  Evaluation of the intrinsic antiviral activity of different doses and dose regimens of JNJ-47910382 in chronic HCV-genotype-1 infected subjects, as measured by the HCV RNA decrease from baseline (Day 1) over time.
Number of participants with adverse events as a measure of safety and tolerability | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (6):
- Germany (6):
  - Hamburg
  - Kiel
  - Mainz
  - Münster
  - Tübingen
  - Ulm